CLINICAL TRIAL: NCT04253938
Title: Evaluation of Feeding Practices in Latin American Infants at a Medical Home in Austin, Texas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Ana M. Avalos, Assistant Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-05-0141
Record Dates: First submitted 2020-01-09; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education (Other): Visit 1 - Parent/Caregiver will complete a questionnaire about breastfeeding/formula feeding practices and food insecurity. The questionnaire includes a nutrition history, asking how much formula is consumed, number of times they are breastfed per day, what types and amounts of solid foods are consumed, and if vitamins and/or iron drops are given (including frequency and amount). After the questionnaire, the participant will be asked to demonstrate how they typically prepare infant formula. Finally, the PI or designee will provide a brief education about appropriate feeding practices as recommended by the AAP. This will include appropriate formula preparation methods, use of juice, introduction of cow's milk and solids, as well as basic nutrition information.
  Visit 2 - If the family returns for a clinic visit again before the child turns 1 year of age, the same procedures as Visit 1 will be performed, including reinforcement of education.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Subjects will be provided education about AAP approved feeding practices for infants 1 to 12 months of age.

SUMMARY:
The purpose of this study is to determine the methods of formula preparation and feeding practices in Latin American households in the first 12 months of life. There is limited published information on the feeding practices of infants in disadvantaged households, and still less information is available regarding disadvantaged Latin American households.

Studies have shown that certain feeding practices such as diluting infant formula, warming bottles in a microwave, or storing partially used bottles in the refrigerator can be dangerous for the infant. Previous pilot data in other states have documented that up to 15-21% of parents dilute infant formula. Motives for doing so included an attempt to avoid infant hunger, save money, or make formula last longer.

DETAILED DESCRIPTION:
The study will include 2 visits, both occurring at the CommUnity Care clinic during the infant's regularly scheduled doctor's visit. Study visits will coincide with the American Academy of Pediatrics' (AAP) recommendations for timing of visits in the first year of life: prior to 2 months of age a baby will be scheduled for 2 visits (usually at 1 and 2 weeks of life), with subsequent well-child visits scheduled for 2, 4, 6, and 9 months of age. The investigators will seek to enroll subjects (Parent/Caregiver of infant less than 1 year of age) when the child attends any visit prior to the 9 month visit so that the investigators can complete both study visits prior to 1 year of age.

Visit 1 - Parent/Caregiver will complete a questionnaire about breastfeeding/formula feeding practices and food insecurity. The questionnaire includes a nutrition history, asking how much formula is consumed, number of times they are breastfed per day, what types and amounts of solid foods are consumed, and if vitamins and/or iron drops are given (including frequency and amount). After the questionnaire, the participant will be asked to demonstrate how they typically prepare infant formula. Finally, the PI or designee will provide a brief education about appropriate feeding practices as recommended by the AAP.

The study will include 2 visits, both occurring at the CommUnity Care clinic during the infant's regularly scheduled doctor's visit. Study visits will coincide with the American Academy of Pediatrics' (AAP) recommendations for timing of visits in the first year of life: prior to 2 months of age a baby will be scheduled for 2 visits (usually at 1 and 2 weeks of life), with subsequent well-child visits scheduled for 2, 4, 6, and 9 months of age. The investigators will seek to enroll subjects (Parent/Caregiver of infant less than 1 year of age) when the child attends any visit prior to the 9 month visit so that the investigators can complete both study visits prior to 1 year of age.

Visit 1 - Parent/Caregiver will complete a questionnaire about breastfeeding/formula feeding practices and food insecurity. The questionnaire includes a nutrition history, asking how much formula is consumed, number of times they are breastfed per day, what types and amounts of solid foods are consumed, and if vitamins and/or iron drops are given (including frequency and amount). After the questionnaire, the participant will be asked to demonstrate how they typically prepare infant formula. Finally, the PI or designee will provide a brief education about appropriate feeding practices as recommended by the AAP. This will include appropriate formula preparation methods, use of juice, introduction of cow's milk and solids, as well as basic nutrition information.

Visit 2 - If the family returns for a clinic visit again before the child turns 1 year of age, the same procedures as Visit 1 will be performed, including reinforcement of education.

The infant's anthropometrics and medical history will be obtained from the EMR.

This pilot data would be the foundation for a larger, more intensive study to determine prevalence of inappropriate feeding strategies among Latin American families and best strategies to educate and inform.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of Latin American infants who are 9 months of age or younger
* Patients at a local CommUnity Care Clinic

Exclusion Criteria:

* Caregivers of Latin American infants over 9 months of age
* Infants who are not Latin American
* Infants with with significant underlying health problems that require feeding modifications such as naso-gastric feedings or concentrated feeds

Ages: 1 Week to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Feeding Score | Up to 1 year
  The investigators will seek to answer the question, "Is there a difference in feeding score between first and second visit" where the feeding score is the sum of points given to 4 inappropriate liquid feeding practices (1. Overdilution of infant formula, 2. Use of sugar water, 3. Cow's milk, and 4. Juice, at 25 points each).

SECONDARY OUTCOMES:
Food insecurity | Up to 1 year
  Food insecurity questionnaire (from a validated short form of the Food Security Scale, Blumberg et al, Am J Public Health, 1999)
Nutrition history | Up to 1 year
  Intake amount and frequency (solid foods, breastfeeding, infant formula), type of infant formula, vitamins and/or iron drops. Feeding practices questions are based on a similar validated survey by Burkhart et al, Clin Pediatri, 2012 and a Perrigo survey from 2018.

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Medical School, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No